CLINICAL TRIAL: NCT03602014
Title: Dose Response to the Norepinephrine Precursor Droxidopa in Hypotensive Individuals With Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Principal Investigator, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEC-17-042
Record Dates: First submitted 2018-02-15; First posted 2018-07-26 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Hypotension, Orthostatic; Hypotension; Spinal Cord Injuries
Keywords: Hypotension; Spinal Cord Injury; Droxidopa; Northera; Neurogenic Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic; Hypotension; Spinal Cord Injuries | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study 1: Dose Optimization of Northera (Experimental): Subjects will be administered oral droxidopa in a dose escalation, open-label manner beginning with 200 mg. The dose will be adjusted upwards by 100 mg on subsequent visits until average Systolic Blood Pressure (SBP) recorded 60-120 minutes after dose administration is 111-139 mmHg in males and 101-139 mmHg in females, sustained elevation (≥ 30 consecutive minutes) in seated SBP ≥ 140/100 mmHg, maximum dose of 800 mg is reached without adequate SBP response. Subjects will visit the testing laboratory on as few as 1 (200 mg) and as many as 7 (800 mg) days. Seated cardiovascular assessments will be monitored and recorded at 15-minute intervals for 4-hours, and the side effects questionnaire will be administered hourly during the 4-hour study. Each study visit will take about 5 hours.
  Interventions: Drug: Northera
- Study 2: Blinded Placebo & Northera (Placebo Comparator): Participants will then be administered either oral optimal dose of Northera (Droxidopa) or matching placebo in a double-blinded manner and will remain in the supine position for 60 minutes. Subjects will remain in their wheelchair for instrumentation, which will include: 1) ECG, 2) brachial BP, 3) finger arteriolar BP and 4) Cerebral Blood Flow velocity (CBFv).
  Interventions: Drug: Northera; Other: Placebo

INTERVENTIONS:
Drug: Northera — Study 1 is a dose optimization, open-label trial of Northera from a dose range of 200mg up to 800mg.
  Other Names: Droxidopa
Other: Placebo — Study 2 is blinded placebo controlled trial using the individualized optimal dose of droxidopa determined by study 1.
  Arms: Study 2: Blinded Placebo & Northera

SUMMARY:
The goal of this study is to determine the efficacy of the drug Droxidopa (Northera) in increasing blood pressure in subject with hypotension, low blood pressure, which is classified as blood pressure less than 110/70 in males and 100/70 in females. The first aim is to determine the proportion of subject with Spinal Cord Injury (SCI) who have a normotensive response to Droxidopa. The second is to determine the proportion of subject with SCI who express a hypertensive response to Droxidopa. A Normal blood pressure ranges from 111-139 in males and 101-139 in females and a hypertensive blood pressure is anything higher than 140 in males and females.

The study would take place in James J. Peters VA Medical Center (JJPVAMC) and The Icahn School of Medicine at Mount Sinai (ISMMS) in Manhattan, New York.

DETAILED DESCRIPTION:
Interruption of sympathetic cardiovascular autonomic regulation following spinal cord injury (SCI) is associated with significantly reduced plasma norepinephrine (NE) levels, hypotension and orthostatic hypotension (OH), particularly in individuals with high cord lesions. Although the incidence of hypotension is reported to be as high as 70% in persons with cervical lesions (i.e., tetraplegia), the vast majority of these individuals remains asymptomatic and, therefore, does not raise clinical concern, or prompt intervention. While it is appreciated that clinicians are faced with substantial challenges in managing blood pressure (BP) in persons with SCI, contrary to the prevailing belief, asymptomatic hypotension and OH are not benign conditions. Reports suggest that asymptomatic hypotensive individuals with SCI may have subclinical cognitive dysfunction affecting memory and attention processing and increased incidence of fatigue and depression compared to normotensive individuals with SCI. It must be appreciated that to date, there are no FDA approved pharmaceutical options proven to be safe and effective for treatment of hypotension and OH in the SCI population. Until 2014, midodrine hydrochloride was the only agent with FDA approval for treatment of symptomatic neurogenic OH (NOH). Midodrine, an alpha-agonist, is the most commonly prescribed agent used to treat symptomatic hypotension in the SCI population despite a lack of convincing evidence of safety or efficacy. In 2014 droxidopa (L-threo-3,4-dihydroxyphenylserine - NORTHERA; Chelsea Therapeutics, Charlotte, NC) was approved by the FDA for treatment of symptomatic NOH based on data collected in conditions of autonomic dysfunction. Droxidopa is a NE precursor that is stored in neuronal and non-neuronal tissue and has been shown to increase standing BP and reduce symptoms of orthostatic intolerance in individuals with symptomatic NOH. We recently reported preliminary evidence of a mean increase in seated BP in individuals with SCI following oral administration of 400 mg of droxidopa; however, this dose was effective in only 5 of the 10 subjects tested and the BP effect waned over a 4-hour observation. Because of its unique pharmacokinetic profile, droxidopa is a highly promising agent to treat hypotension in persons with SCI. As such; there exists a pressing imperative to determine the clinical value and safety of droxidopa in hypotensive individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

Study 1:

1. Male or Female, age 18 to 89 with traumatic SCI.
2. SCI Subjects (n=40):

   1. Any level of injury;
   2. Any American Spinal Injury Association Impairment Scale (AIS) grade of SCI;
   3. Non-ventilator dependent
   4. Primarily wheelchair dependent for mobility;
   5. Duration of injury < 1 year
3. Low Blood Pressure:

   1. Systolic BP less than 110 mmHg and/or diastolic BP less than 70 mmHg for males.
   2. Systolic BP less than 100 mmHg and/or diastolic BP less than 70 mmHg for females.
4. Primary Language is English.
5. Able to provide informed consent

   Study 2:
6. Male or Female, age 18 to 89 with traumatic SCI.
7. SCI Subjects (n=40):

   1. Any level of injury;
   2. Any AIS grade of SCI;
   3. Non-ventilator dependent
   4. Primarily wheelchair dependent for mobility
   5. Duration of injury < 1 year
8. Low Blood Pressure:

   1. Systolic BP less than 110 mmHg and/or diastolic BP less than 70 mmHg for males.
   2. Systolic BP less than 100 mmHg and/or diastolic BP less than 70 mmHg for females.
9. Primary Language is English.
10. Able to provide informed consent
11. Showed a normotensive blood pressure in response to Droxidopa during study 1.

Exclusion Criteria:

* Current illness or infection
* Individuals with frequent or severe autonomic dysreflexia:

  1. More than 3 symptomatic events per week
  2. BP ≥140/90 mmHg
  3. Significant adverse subjective symptoms reporting
* Hypertension
* Any neurological condition other than SCI (Alzheimer's disease, dementia, stroke, multiple sclerosis, Parkinson's disease, etc.)
* History of epilepsy or other seizure disorder
* History of traumatic brain injury (TBI)
* Liver or kidney disease
* Bladder problems including blockage of the urine and/or weak urine stream.
* Diagnosis of a psychiatric disorder such as schizophrenia or bipolar disorder
* Known artery disease, heart failure, Atrio-ventricular block, and irregular heartbeat
* Any allergies to droxidopa, asprin, polyethylene oxide, polyethylene glycol, hydroxypropyl cellulose, butylated hydroxytoluene, magnesium stearate, hypromellose, yellow ferric oxide, and red ferric oxide
* Major surgery in the last 30 days
* Illicit drug abuse in the past 6 months
* Pregnant
* Your prescription medications will be reviewed by the study investigators and research staff. If you are currently taking medications to treat any of the following please make the investigators aware:

  d. Depression, Schizophrenia, Attention Deficit Hyperactivity Disorder (ADHD) e. Pain (opioids) f. Infection or illness (antibiotics) g. Erectile dysfunction (Viagra, Cialis, etc.) h. Overactive bladder i. High or low blood pressure j. Migraine headaches k. Malaria l. asthma

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, Ed.D, Principal Investigator — James J. Peter's VAMC
Locations (2):
- United States (2):
  - The Icahn School of Medicine at Mount Sinai, New York, New York
  - James J. Peters Veteran's Affair Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claydon VE, Krassioukov AV. Orthostatic hypotension and autonomic pathways after spinal cord injury. J Neurotrauma. 2006 Dec;23(12):1713-25. doi: 10.1089/neu.2006.23.1713. PMID 17184183
- [Background] GUTTMANN L, MUNRO AF, ROBINSON R, WALSH JJ. EFFECT OF TILTING ON THE CARDIOVASCULAR RESPONSES AND PLASMA CATECHOLAMINE LEVELS IN SPINAL MAN. Paraplegia. 1963 May;1:4-18. doi: 10.1038/sc.1963.2. No abstract available. PMID 14087938
- [Background] Mathias CJ, Christensen NJ, Corbett JL, Frankel HL, Goodwin TJ, Peart WS. Plasma catecholamines, plasma renin activity and plasma aldosterone in tetraplegic man, horizontal and tilted. Clin Sci Mol Med. 1975 Oct;49(4):291-9. doi: 10.1042/cs0490291. PMID 1192688
- [Background] Wecht JM, Weir JP, Goldstein DS, Krothe-Petroff A, Spungen AM, Holmes C, Bauman WA. Direct and reflexive effects of nitric oxide synthase inhibition on blood pressure. Am J Physiol Heart Circ Physiol. 2008 Jan;294(1):H190-7. doi: 10.1152/ajpheart.00366.2007. Epub 2007 Oct 26. PMID 17965289
- [Background] Wecht JM, Zhu C, Weir JP, Yen C, Renzi C, Galea M. A prospective report on the prevalence of heart rate and blood pressure abnormalities in veterans with spinal cord injuries. J Spinal Cord Med. 2013 Sep;36(5):454-62. doi: 10.1179/2045772313Y.0000000109. PMID 23941793
- [Background] Zhu C, Galea M, Livote E, Signor D, Wecht JM. A retrospective chart review of heart rate and blood pressure abnormalities in veterans with spinal cord injury. J Spinal Cord Med. 2013 Sep;36(5):463-75. doi: 10.1179/2045772313Y.0000000145. PMID 23941794
- [Background] Jegede AB, Rosado-Rivera D, Bauman WA, Cardozo CP, Sano M, Moyer JM, Brooks M, Wecht JM. Cognitive performance in hypotensive persons with spinal cord injury. Clin Auton Res. 2010 Feb;20(1):3-9. doi: 10.1007/s10286-009-0036-z. Epub 2009 Oct 16. PMID 19842013
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Perturbed and spontaneous regional cerebral blood flow responses to changes in blood pressure after high-level spinal cord injury: the effect of midodrine. J Appl Physiol (1985). 2014 Mar 15;116(6):645-53. doi: 10.1152/japplphysiol.01090.2013. Epub 2014 Jan 16. PMID 24436297
- [Background] Phillips AA, Warburton DE, Ainslie PN, Krassioukov AV. Regional neurovascular coupling and cognitive performance in those with low blood pressure secondary to high-level spinal cord injury: improved by alpha-1 agonist midodrine hydrochloride. J Cereb Blood Flow Metab. 2014 May;34(5):794-801. doi: 10.1038/jcbfm.2014.3. Epub 2014 Jan 29. PMID 24473484
- [Background] Wecht JM, Bauman WA. Decentralized cardiovascular autonomic control and cognitive deficits in persons with spinal cord injury. J Spinal Cord Med. 2013 Mar;36(2):74-81. doi: 10.1179/2045772312Y.0000000056. PMID 23809520
- [Background] Wecht JM, Rosado-Rivera D, Jegede A, Cirnigliaro CM, Jensen MA, Kirshblum S, Bauman WA. Systemic and cerebral hemodynamics during cognitive testing. Clin Auton Res. 2012 Feb;22(1):25-33. doi: 10.1007/s10286-011-0139-1. Epub 2011 Jul 27. PMID 21792728
- [Background] Krassioukov A, Eng JJ, Warburton DE, Teasell R; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2009 May;90(5):876-85. doi: 10.1016/j.apmr.2009.01.009. PMID 19406310
- [Background] Kaufmann H, Freeman R, Biaggioni I, Low P, Pedder S, Hewitt LA, Mauney J, Feirtag M, Mathias CJ; NOH301 Investigators. Droxidopa for neurogenic orthostatic hypotension: a randomized, placebo-controlled, phase 3 trial. Neurology. 2014 Jul 22;83(4):328-35. doi: 10.1212/WNL.0000000000000615. Epub 2014 Jun 18. PMID 24944260
- [Background] Kaufmann H, Norcliffe-Kaufmann L, Palma JA. Droxidopa in neurogenic orthostatic hypotension. Expert Rev Cardiovasc Ther. 2015;13(8):875-91. doi: 10.1586/14779072.2015.1057504. Epub 2015 Jun 19. PMID 26092297
- [Background] Kaufmann H, Saadia D, Voustianiouk A, Goldstein DS, Holmes C, Yahr MD, Nardin R, Freeman R. Norepinephrine precursor therapy in neurogenic orthostatic hypotension. Circulation. 2003 Aug 12;108(6):724-8. doi: 10.1161/01.CIR.0000083721.49847.D7. Epub 2003 Jul 28. PMID 12885750
- [Background] Wecht JM, Rosado-Rivera D, Weir JP, Ivan A, Yen C, Bauman WA. Hemodynamic effects of L-threo-3,4-dihydroxyphenylserine (Droxidopa) in hypotensive individuals with spinal cord injury. Arch Phys Med Rehabil. 2013 Oct;94(10):2006-12. doi: 10.1016/j.apmr.2013.03.028. Epub 2013 Apr 18. PMID 23602882
- [Background] Goldstein DS, Holmes C, Kaufmann H, Freeman R. Clinical pharmacokinetics of the norepinephrine precursor L-threo-DOPS in primary chronic autonomic failure. Clin Auton Res. 2004 Dec;14(6):363-8. doi: 10.1007/s10286-004-0221-z. PMID 15666063
- [Background] Carlozzi NE, Fyffe D, Morin KG, Byrne R, Tulsky DS, Victorson D, Lai JS, Wecht JM. Impact of blood pressure dysregulation on health-related quality of life in persons with spinal cord injury: development of a conceptual model. Arch Phys Med Rehabil. 2013 Sep;94(9):1721-30. doi: 10.1016/j.apmr.2013.02.024. Epub 2013 Mar 14. PMID 23499779
- [Background] Dolinak D, Balraj E. Autonomic dysreflexia and sudden death in people with traumatic spinal cord injury. Am J Forensic Med Pathol. 2007 Jun;28(2):95-8. doi: 10.1097/PAF.0b013e3180600f99. PMID 17525555
- [Background] Courtois FJ, Charvier KF, Leriche A, Vezina JG, Cote M, Belanger M. Blood pressure changes during sexual stimulation, ejaculation and midodrine treatment in men with spinal cord injury. BJU Int. 2008 Feb;101(3):331-7. doi: 10.1111/j.1464-410X.2007.07254.x. Epub 2007 Oct 8. PMID 17922856
- [Background] Barber DB, Rogers SJ, Fredrickson MD, Able AC. Midodrine hydrochloride and the treatment of orthostatic hypotension in tetraplegia: two cases and a review of the literature. Spinal Cord. 2000 Feb;38(2):109-11. doi: 10.1038/sj.sc.3100959. PMID 10762185
- [Background] Mukand J, Karlin L, Barrs K, Lublin P. Midodrine for the management of orthostatic hypotension in patients with spinal cord injury: A case report. Arch Phys Med Rehabil. 2001 May;82(5):694-6. doi: 10.1053/apmr.2001.22350. PMID 11346851
- [Background] Canosa-Hermida E, Mondelo-Garcia C, Ferreiro-Velasco ME, Salvador-de la Barrera S, Montoto-Marques A, Rodriguez-Sotillo A, Vizoso-Hermida JR. Refractory orthostatic hypotension in a patient with a spinal cord injury: Treatment with droxidopa. J Spinal Cord Med. 2018 Jan;41(1):115-118. doi: 10.1080/10790268.2016.1274093. Epub 2017 Jan 24. PMID 28114866
- [Background] Nieshoff EC, Birk TJ, Birk CA, Hinderer SR, Yavuzer G. Double-blinded, placebo-controlled trial of midodrine for exercise performance enhancement in tetraplegia: a pilot study. J Spinal Cord Med. 2004;27(3):219-25. doi: 10.1080/10790268.2004.11753752. PMID 15478524
- [Background] Wecht JM, Rosado-Rivera D, Handrakis JP, Radulovic M, Bauman WA. Effects of midodrine hydrochloride on blood pressure and cerebral blood flow during orthostasis in persons with chronic tetraplegia. Arch Phys Med Rehabil. 2010 Sep;91(9):1429-35. doi: 10.1016/j.apmr.2010.06.017. PMID 20801263
- [Background] Muneta S, Iwata T, Hiwada K, Murakami E, Sato Y, Imamura Y. Effect of L-threo-3, 4-dihydroxyphenylserine on orthostatic hypotension in a patient with spinal cord injury. Jpn Circ J. 1992 Mar;56(3):243-7. doi: 10.1253/jcj.56.243. PMID 1552652
- [Background] Kannel WB, Wolf PA, Verter J, McNamara PM. Epidemiologic assessment of the role of blood pressure in stroke. The Framingham study. JAMA. 1970 Oct 12;214(2):301-10. No abstract available. PMID 5469068
- [Background] Robbins JM, Korda H, Shapiro MF. Treatment for a nondisease: the case of low blood pressure. Soc Sci Med. 1982;16(1):27-33. doi: 10.1016/0277-9536(82)90420-8. PMID 7100954
- [Background] MEADOR CK. THE ART AND SCIENCE OF NONDISEASE. N Engl J Med. 1965 Jan 14;272:92-5. doi: 10.1056/NEJM196501142720208. No abstract available. PMID 14223129
- [Background] Barrett-Connor E, Palinkas LA. Low blood pressure and depression in older men: a population based study. BMJ. 1994 Feb 12;308(6926):446-9. doi: 10.1136/bmj.308.6926.446. PMID 8124175
- [Background] Pilgrim JA, Stansfeld S, Marmot M. Low blood pressure, low mood? BMJ. 1992 Jan 11;304(6819):75-8. doi: 10.1136/bmj.304.6819.75. PMID 1737142
- [Background] Rosengren A, Tibblin G, Wilhelmsen L. Low systolic blood pressure and self perceived wellbeing in middle aged men. BMJ. 1993 Jan 23;306(6872):243-6. doi: 10.1136/bmj.306.6872.243. PMID 8443523
- [Background] Wessely S, Nickson J, Cox B. Symptoms of low blood pressure: a population study. BMJ. 1990 Aug 18-25;301(6748):362-5. doi: 10.1136/bmj.301.6748.362. PMID 2400856
- [Background] Niu K, Hozawa A, Awata S, Guo H, Kuriyama S, Seki T, Ohmori-Matsuda K, Nakaya N, Ebihara S, Wang Y, Tsuji I, Nagatomi R. Home blood pressure is associated with depressive symptoms in an elderly population aged 70 years and over: a population-based, cross-sectional analysis. Hypertens Res. 2008 Mar;31(3):409-16. doi: 10.1291/hypres.31.409. PMID 18497459
- [Background] Hildrum B, Mykletun A, Holmen J, Dahl AA. Effect of anxiety and depression on blood pressure: 11-year longitudinal population study. Br J Psychiatry. 2008 Aug;193(2):108-13. doi: 10.1192/bjp.bp.107.045013. PMID 18669991
- [Background] Hildrum B, Mykletun A, Stordal E, Bjelland I, Dahl AA, Holmen J. Association of low blood pressure with anxiety and depression: the Nord-Trondelag Health Study. J Epidemiol Community Health. 2007 Jan;61(1):53-8. doi: 10.1136/jech.2005.044966. PMID 17183016
- [Background] Jorm AF. Association of hypotension with positive and negative affect and depressive symptoms in the elderly. Br J Psychiatry. 2001 Jun;178:553-5. doi: 10.1192/bjp.178.6.553. PMID 11388973
- [Background] Kim BS, Bae JN, Cho MJ. Depressive symptoms in elderly adults with hypotension: different associations with positive and negative affect. J Affect Disord. 2010 Dec;127(1-3):359-64. doi: 10.1016/j.jad.2010.06.024. PMID 20619901
- [Background] Paterniti S, Verdier-Taillefer MH, Geneste C, Bisserbe JC, Alperovitch A. Low blood pressure and risk of depression in the elderly. A prospective community-based study. Br J Psychiatry. 2000 May;176:464-7. doi: 10.1192/bjp.176.5.464. PMID 10912223
- [Background] Stroup-Benham CA, Markides KS, Black SA, Goodwin JS. Relationship between low blood pressure and depressive symptomatology in older people. J Am Geriatr Soc. 2000 Mar;48(3):250-5. doi: 10.1111/j.1532-5415.2000.tb02642.x. PMID 10733049
- [Background] Donner-Banzhoff N, Chan Y, Szalai JP, Hilditch JR. Low blood pressure associated with low mood: a red herring? J Clin Epidemiol. 1997 Oct;50(10):1175-81. doi: 10.1016/s0895-4356(97)00157-1. PMID 9368526
- [Background] Herva A, Rasanen P, Miettunen J, Timonen M, Laksy K, Veijola J, Laitinen J, Ruokonen A, Joukamaa M. Co-occurrence of metabolic syndrome with depression and anxiety in young adults: the Northern Finland 1966 Birth Cohort Study. Psychosom Med. 2006 Mar-Apr;68(2):213-6. doi: 10.1097/01.psy.0000203172.02305.ea. PMID 16554385
- [Background] Fann JR, Bombardier CH, Richards JS, Tate DG, Wilson CS, Temkin N; PRISMS Investigators. Depression after spinal cord injury: comorbidities, mental health service use, and adequacy of treatment. Arch Phys Med Rehabil. 2011 Mar;92(3):352-60. doi: 10.1016/j.apmr.2010.05.016. Epub 2011 Jan 20. PMID 21255766
- [Background] Hoffman JM, Bombardier CH, Graves DE, Kalpakjian CZ, Krause JS. A longitudinal study of depression from 1 to 5 years after spinal cord injury. Arch Phys Med Rehabil. 2011 Mar;92(3):411-8. doi: 10.1016/j.apmr.2010.10.036. PMID 21353823
- [Background] Davidoff G, Roth E, Thomas P, Doljanac R, Dijkers M, Berent S, Morris J, Yarkony G. Depression and neuropsychological test performance in acute spinal cord injury patients: lack of correlation. Arch Clin Neuropsychol. 1990;5(1):77-88. PMID 14589546
- [Background] Wecht JM, Weir JP, Martinez S, Eraifej M, Bauman WA. Orthostatic hypotension and orthostatic hypertension in American veterans. Clin Auton Res. 2016 Feb;26(1):49-58. doi: 10.1007/s10286-015-0328-4. Epub 2015 Dec 22. PMID 26695397
- [Background] Yap PL, Niti M, Yap KB, Ng TP. Orthostatic hypotension, hypotension and cognitive status: early comorbid markers of primary dementia? Dement Geriatr Cogn Disord. 2008;26(3):239-46. doi: 10.1159/000160955. Epub 2008 Oct 8. PMID 18841007
- [Background] Launer LJ, Masaki K, Petrovitch H, Foley D, Havlik RJ. The association between midlife blood pressure levels and late-life cognitive function. The Honolulu-Asia Aging Study. JAMA. 1995 Dec 20;274(23):1846-51. PMID 7500533
- [Background] Weisz N, Schandry R, Jacobs AM, Mialet JP, Duschek S. Early contingent negative variation of the EEG and attentional flexibility are reduced in hypotension. Int J Psychophysiol. 2002 Sep;45(3):253-60. doi: 10.1016/s0167-8760(02)00032-6. PMID 12208532
- [Background] Duschek S, Schandry R. Cognitive performance and cerebral blood flow in essential hypotension. Psychophysiology. 2004 Nov;41(6):905-13. doi: 10.1111/j.1469-8986.2004.00249.x. PMID 15563343
- [Background] Duschek S, Matthias E, Schandry R. Essential hypotension is accompanied by deficits in attention and working memory. Behav Med. 2005 Winter;30(4):149-58. doi: 10.3200/BMED.30.4.149-160. PMID 15981893
- [Background] Frewen J, Finucane C, Savva GM, Boyle G, Kenny RA. Orthostatic hypotension is associated with lower cognitive performance in adults aged 50 plus with supine hypertension. J Gerontol A Biol Sci Med Sci. 2014 Jul;69(7):878-85. doi: 10.1093/gerona/glt171. Epub 2013 Nov 8. PMID 24214492
- [Background] Frewen J, Savva GM, Boyle G, Finucane C, Kenny RA. Cognitive performance in orthostatic hypotension: findings from a nationally representative sample. J Am Geriatr Soc. 2014 Jan;62(1):117-22. doi: 10.1111/jgs.12592. PMID 25180380
- [Background] Mehrabian S, Duron E, Labouree F, Rollot F, Bune A, Traykov L, Hanon O. Relationship between orthostatic hypotension and cognitive impairment in the elderly. J Neurol Sci. 2010 Dec 15;299(1-2):45-8. doi: 10.1016/j.jns.2010.08.056. Epub 2010 Sep 19. PMID 20855089
- [Background] Sambati L, Calandra-Buonaura G, Poda R, Guaraldi P, Cortelli P. Orthostatic hypotension and cognitive impairment: a dangerous association? Neurol Sci. 2014 Jun;35(6):951-7. doi: 10.1007/s10072-014-1686-8. Epub 2014 Mar 4. PMID 24590841
- [Background] Rose KM, Couper D, Eigenbrodt ML, Mosley TH, Sharrett AR, Gottesman RF. Orthostatic hypotension and cognitive function: the Atherosclerosis Risk in Communities Study. Neuroepidemiology. 2010;34(1):1-7. doi: 10.1159/000255459. Epub 2009 Nov 5. PMID 19893322
- [Background] Duschek S, Hadjamu M, Schandry R. Enhancement of cerebral blood flow and cognitive performance following pharmacological blood pressure elevation in chronic hypotension. Psychophysiology. 2007 Jan;44(1):145-53. doi: 10.1111/j.1469-8986.2006.00472.x. PMID 17241150
- [Background] Duschek S, Hadjamu M, Schandry R. Dissociation between cortical activation and cognitive performance under pharmacological blood pressure elevation in chronic hypotension. Biol Psychol. 2007 Jul;75(3):277-85. doi: 10.1016/j.biopsycho.2007.03.007. Epub 2007 Apr 5. PMID 17481800
- [Background] Hillis AE, Ulatowski JA, Barker PB, Torbey M, Ziai W, Beauchamp NJ, Oh S, Wityk RJ. A pilot randomized trial of induced blood pressure elevation: effects on function and focal perfusion in acute and subacute stroke. Cerebrovasc Dis. 2003;16(3):236-46. doi: 10.1159/000071122. PMID 12865611
- [Background] Wecht JM, Weir JP, Radulovic M, Bauman WA. Effects of midodrine and L-NAME on systemic and cerebral hemodynamics during cognitive activation in spinal cord injury and intact controls. Physiol Rep. 2016 Feb;4(3):e12683. doi: 10.14814/phy2.12683. PMID 26869679
- [Background] Wecht JM, Radulovic M, Rosado-Rivera D, Zhang RL, LaFountaine MF, Bauman WA. Orthostatic effects of midodrine versus L-NAME on cerebral blood flow and the renin-angiotensin-aldosterone system in tetraplegia. Arch Phys Med Rehabil. 2011 Nov;92(11):1789-95. doi: 10.1016/j.apmr.2011.03.022. Epub 2011 Jul 16. PMID 21762873
- [Background] Pemberton J. Does constitutional hypotension exist? BMJ. 1989 Mar 11;298(6674):660-2. doi: 10.1136/bmj.298.6674.660. No abstract available. PMID 2496798
- [Background] Shapiro MF, Korda H, Robbins J. Diagnosis and treatment of low blood pressure in a Canadian community. Can Med Assoc J. 1982 Apr 15;126(8):918-20. PMID 20313723
- [Background] Arterial hypertension. Report of a WHO expert committee. World Health Organ Tech Rep Ser. 1978;(628):7-56. No abstract available. PMID 103326
- [Background] Lindholm L, Lanke J, Bengtsson B, Ejlertsson G, Thulin T, Schersten B. Both high and low blood pressures risk indicators of death in middle-aged males. Isotonic regression of blood pressure on age applied to data from a 13-year prospective study. Acta Med Scand. 1985;218(5):473-80. doi: 10.1111/j.0954-6820.1985.tb08876.x. PMID 4091047
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. The Consensus Committee of the American Autonomic Society and the American Academy of Neurology. Neurology. 1996 May;46(5):1470. doi: 10.1212/wnl.46.5.1470. No abstract available. PMID 8628505
- [Background] Wu JS, Yang YC, Lu FH, Wu CH, Chang CJ. Population-based study on the prevalence and correlates of orthostatic hypotension/hypertension and orthostatic dizziness. Hypertens Res. 2008 May;31(5):897-904. doi: 10.1291/hypres.31.897. PMID 18712045
- [Background] Rose KM, Eigenbrodt ML, Biga RL, Couper DJ, Light KC, Sharrett AR, Heiss G. Orthostatic hypotension predicts mortality in middle-aged adults: the Atherosclerosis Risk In Communities (ARIC) Study. Circulation. 2006 Aug 15;114(7):630-6. doi: 10.1161/CIRCULATIONAHA.105.598722. Epub 2006 Aug 7. PMID 16894039
- [Background] Rutan GH, Hermanson B, Bild DE, Kittner SJ, LaBaw F, Tell GS. Orthostatic hypotension in older adults. The Cardiovascular Health Study. CHS Collaborative Research Group. Hypertension. 1992 Jun;19(6 Pt 1):508-19. doi: 10.1161/01.hyp.19.6.508. PMID 1592445
- [Background] Shibao C, Grijalva CG, Raj SR, Biaggioni I, Griffin MR. Orthostatic hypotension-related hospitalizations in the United States. Am J Med. 2007 Nov;120(11):975-80. doi: 10.1016/j.amjmed.2007.05.009. PMID 17976425
- [Background] Eigenbrodt ML, Rose KM, Couper DJ, Arnett DK, Smith R, Jones D. Orthostatic hypotension as a risk factor for stroke: the atherosclerosis risk in communities (ARIC) study, 1987-1996. Stroke. 2000 Oct;31(10):2307-13. doi: 10.1161/01.str.31.10.2307. PMID 11022055
- [Background] Rose KM, Tyroler HA, Nardo CJ, Arnett DK, Light KC, Rosamond W, Sharrett AR, Szklo M. Orthostatic hypotension and the incidence of coronary heart disease: the Atherosclerosis Risk in Communities study. Am J Hypertens. 2000 Jun;13(6 Pt 1):571-8. doi: 10.1016/s0895-7061(99)00257-5. PMID 10912737
- [Background] Masaki KH, Schatz IJ, Burchfiel CM, Sharp DS, Chiu D, Foley D, Curb JD. Orthostatic hypotension predicts mortality in elderly men: the Honolulu Heart Program. Circulation. 1998 Nov 24;98(21):2290-5. doi: 10.1161/01.cir.98.21.2290. PMID 9826316
- [Background] Schatz IJ. Orthostatic hypotension predicts mortality. Lessons from the Honolulu Heart Program. Clin Auton Res. 2002 Aug;12(4):223-4. doi: 10.1007/s10286-002-0047-5. No abstract available. PMID 12357271
- [Background] Fedorowski A, Stavenow L, Hedblad B, Berglund G, Nilsson PM, Melander O. Orthostatic hypotension predicts all-cause mortality and coronary events in middle-aged individuals (The Malmo Preventive Project). Eur Heart J. 2010 Jan;31(1):85-91. doi: 10.1093/eurheartj/ehp329. Epub 2009 Aug 20. PMID 19696189
- [Background] Goswami R, Krishan K, Suryaprakash B, Vaidyanathan S, Rao K, Rao MS, Goswami AK, Goel AK, Sharma PL. Circadian desynchronization in pulse rate, systolic and diastolic blood pressure, rectal temperature and urine output in traumatic tetraplegics. Indian J Physiol Pharmacol. 1985 Oct-Dec;29(4):199-206. PMID 3842372
- [Background] Krum H, Louis WJ, Brown DJ, Jackman GP, Howes LG. Diurnal blood pressure variation in quadriplegic chronic spinal cord injury patients. Clin Sci (Lond). 1991 Mar;80(3):271-6. doi: 10.1042/cs0800271. PMID 1850688
- [Background] Munakata M, Kameyama J, Kanazawa M, Nunokawa T, Moriai N, Yoshinaga K. Circadian blood pressure rhythm in patients with higher and lower spinal cord injury: simultaneous evaluation of autonomic nervous activity and physical activity. J Hypertens. 1997 Dec;15(12 Pt 2):1745-9. doi: 10.1097/00004872-199715120-00083. PMID 9488233
- [Background] Krassioukov AV, Karlsson AK, Wecht JM, Wuermser LA, Mathias CJ, Marino RJ; Joint Committee of American Spinal Injury Association and International Spinal Cord Society. Assessment of autonomic dysfunction following spinal cord injury: rationale for additions to International Standards for Neurological Assessment. J Rehabil Res Dev. 2007;44(1):103-12. doi: 10.1682/jrrd.2005.10.0159. PMID 17551864
- [Background] Frankel HL, Michaelis LS, Golding DR, Beral V. The blood pressure in paraplegia. I. Paraplegia. 1972 Nov;10(3):193-200. doi: 10.1038/sc.1972.32. No abstract available. PMID 4636920
- [Background] Lehmann KG, Lane JG, Piepmeier JM, Batsford WP. Cardiovascular abnormalities accompanying acute spinal cord injury in humans: incidence, time course and severity. J Am Coll Cardiol. 1987 Jul;10(1):46-52. doi: 10.1016/s0735-1097(87)80158-4. PMID 3597994
- [Background] Teasell RW, Arnold JM, Krassioukov A, Delaney GA. Cardiovascular consequences of loss of supraspinal control of the sympathetic nervous system after spinal cord injury. Arch Phys Med Rehabil. 2000 Apr;81(4):506-16. doi: 10.1053/mr.2000.3848. PMID 10768544
- [Background] Blackmer J. Orthostatic hypotension in spinal cord injured patients. J Spinal Cord Med. 1997 Apr;20(2):212-7. doi: 10.1080/10790268.1997.11719471. PMID 9144611
- [Background] Claydon VE, Steeves JD, Krassioukov A. Orthostatic hypotension following spinal cord injury: understanding clinical pathophysiology. Spinal Cord. 2006 Jun;44(6):341-51. doi: 10.1038/sj.sc.3101855. Epub 2005 Nov 22. PMID 16304564
- [Background] Illman A, Stiller K, Williams M. The prevalence of orthostatic hypotension during physiotherapy treatment in patients with an acute spinal cord injury. Spinal Cord. 2000 Dec;38(12):741-7. doi: 10.1038/sj.sc.3101089. PMID 11175374
- [Background] Lopes P, Figoni S. Current literature on orthostatic hypotension and training in SCI patients. Am Correct Ther J. 1982 Mar-Apr;36(2):56-9. No abstract available. PMID 7048872
- [Background] Ekland MB, Krassioukov AV, McBride KE, Elliott SL. Incidence of autonomic dysreflexia and silent autonomic dysreflexia in men with spinal cord injury undergoing sperm retrieval: implications for clinical practice. J Spinal Cord Med. 2008;31(1):33-9. doi: 10.1080/10790268.2008.11753978. PMID 18533409
- [Background] Wecht JM, Weir JP, Galea M, Martinez S, Bauman WA. Prevalence of abnormal systemic hemodynamics in veterans with and without spinal cord injury. Arch Phys Med Rehabil. 2015 Jun;96(6):1071-9. doi: 10.1016/j.apmr.2015.01.018. Epub 2015 Feb 4. PMID 25660005
- [Background] Wecht JM, Radulovic M, Weir JP, Lessey J, Spungen AM, Bauman WA. Partial angiotensin-converting enzyme inhibition during acute orthostatic stress in persons with tetraplegia. J Spinal Cord Med. 2005;28(2):103-8. doi: 10.1080/10790268.2005.11753806. PMID 15889697
- [Background] West CR, Squair JW, McCracken L, Currie KD, Somvanshi R, Yuen V, Phillips AA, Kumar U, McNeill JH, Krassioukov AV. Cardiac Consequences of Autonomic Dysreflexia in Spinal Cord Injury. Hypertension. 2016 Nov;68(5):1281-1289. doi: 10.1161/HYPERTENSIONAHA.116.07919. Epub 2016 Oct 3. PMID 27698067
- [Background] Wecht JM, De Meersman RE, Weir JP, Spungen AM, Bauman WA. Cardiac autonomic responses to progressive head-up tilt in individuals with paraplegia. Clin Auton Res. 2003 Dec;13(6):433-8. doi: 10.1007/s10286-003-0115-5. PMID 14673693
- [Background] Phillips AA, Ainslie PN, Warburton DE, Krassioukov AV. Cerebral Blood Flow Responses to Autonomic Dysreflexia in Humans with Spinal Cord Injury. J Neurotrauma. 2016 Feb 1;33(3):315-8. doi: 10.1089/neu.2015.3871. Epub 2016 Jan 7. PMID 26077616
- [Background] Clayton KS, Chubon RA. Factors associated with the quality of life of long-term spinal cord injured persons. Arch Phys Med Rehabil. 1994 Jun;75(6):633-8. doi: 10.1016/0003-9993(94)90184-8. PMID 8002760
- [Background] Fuhrer MJ, Rintala DH, Hart KA, Clearman R, Young ME. Relationship of life satisfaction to impairment, disability, and handicap among persons with spinal cord injury living in the community. Arch Phys Med Rehabil. 1992 Jun;73(6):552-7. PMID 1622304
- [Background] Krassioukov A. Autonomic dysreflexia: current evidence related to unstable arterial blood pressure control among athletes with spinal cord injury. Clin J Sport Med. 2012 Jan;22(1):39-45. doi: 10.1097/JSM.0b013e3182420699. PMID 22222591
- [Background] Krassioukov AV, Furlan JC, Fehlings MG. Autonomic dysreflexia in acute spinal cord injury: an under-recognized clinical entity. J Neurotrauma. 2003 Aug;20(8):707-16. doi: 10.1089/089771503767869944. PMID 12965050
- [Background] Yokomizo Y, Goubara A, Tanaka K, Yokoyama O. [A case of cerebellar hemorrhage secondary to autonomic dysreflexia (AD) in a patient with cervical spinal cord injury]. Hinyokika Kiyo. 2010 Nov;56(11):659-61. Japanese. PMID 21187714
- [Background] Eker A, Yigitoglu PH, Ipekdal HI, Tosun A. Acute Onset of Intracerebral Hemorrhage due to Autonomic Dysreflexia. J Korean Neurosurg Soc. 2014 May;55(5):277-9. doi: 10.3340/jkns.2014.55.5.277. Epub 2014 May 31. PMID 25132935
- [Background] Wan D, Krassioukov AV. Life-threatening outcomes associated with autonomic dysreflexia: a clinical review. J Spinal Cord Med. 2014 Jan;37(1):2-10. doi: 10.1179/2045772313Y.0000000098. Epub 2013 Nov 26. PMID 24090418
- [Background] Senard JM, Arias A, Berlan M, Tran MA, Rascol A, Montastruc JL. Pharmacological evidence of alpha 1- and alpha 2-adrenergic supersensitivity in orthostatic hypotension due to spinal cord injury: a case report. Eur J Clin Pharmacol. 1991;41(6):593-6. doi: 10.1007/BF00314991. PMID 1726151
- [Background] Wecht JM, Weir JP, Krothe AH, Spungen AM, Bauman WA. Normalization of supine blood pressure after nitric oxide synthase inhibition in persons with tetraplegia. J Spinal Cord Med. 2007;30(1):5-9. doi: 10.1080/10790268.2007.11753907. PMID 17385265
- [Background] Wecht JM, Radulovic M, Lafountaine MF, Rosado-Rivera D, Zhang RL, Bauman WA. Orthostatic responses to nitric oxide synthase inhibition in persons with tetraplegia. Arch Phys Med Rehabil. 2009 Aug;90(8):1428-34. doi: 10.1016/j.apmr.2009.02.004. PMID 19651280
- [Background] Yamamoto T, Sakakibara R, Yamanaka Y, Uchiyama T, Asahina M, Liu Z, Ito T, Koyama Y, Awa Y, Yamamoto K, Kinou M, Hattori T. Pyridostigmine in autonomic failure: can we treat postural hypotension and bladder dysfunction with one drug? Clin Auton Res. 2006 Aug;16(4):296-8. doi: 10.1007/s10286-006-0358-z. Epub 2006 Jun 21. PMID 16862395
- [Background] Singer W, Sandroni P, Opfer-Gehrking TL, Suarez GA, Klein CM, Hines S, O'Brien PC, Slezak J, Low PA. Pyridostigmine treatment trial in neurogenic orthostatic hypotension. Arch Neurol. 2006 Apr;63(4):513-8. doi: 10.1001/archneur.63.4.noc50340. Epub 2006 Feb 13. PMID 16476804
- [Background] Singer W, Opfer-Gehrking TL, Nickander KK, Hines SM, Low PA. Acetylcholinesterase inhibition in patients with orthostatic intolerance. J Clin Neurophysiol. 2006 Oct;23(5):476-81. doi: 10.1097/01.wnp.0000229946.01494.4c. PMID 17016160
- [Background] Provitera V, Nolano M, Pagano A. Acetylcholinesterase inhibition and orthostatic hypotension. Clin Auton Res. 2006 Apr;16(2):136. doi: 10.1007/s10286-006-0336-5. No abstract available. PMID 16572351
- [Background] Wecht JM, Cirnigliaro CM, Azarelo F, Bauman WA, Kirshblum SC. Orthostatic responses to anticholinesterase inhibition in spinal cord injury. Clin Auton Res. 2015 Jun;25(3):179-87. doi: 10.1007/s10286-015-0272-3. Epub 2015 Apr 28. PMID 25916633
- [Background] Kaufmann H. L-dihydroxyphenylserine (Droxidopa): a new therapy for neurogenic orthostatic hypotension: the US experience. Clin Auton Res. 2008 Mar;18 Suppl 1:19-24. doi: 10.1007/s10286-007-1002-2. Epub 2008 Mar 27. PMID 18368303
- [Background] Mathias CJ. L-dihydroxyphenylserine (Droxidopa) in the treatment of orthostatic hypotension: the European experience. Clin Auton Res. 2008 Mar;18 Suppl 1:25-9. doi: 10.1007/s10286-007-1005-z. Epub 2008 Mar 27. PMID 18368304
- [Background] Isaacson SH, Skettini J. Neurogenic orthostatic hypotension in Parkinson's disease: evaluation, management, and emerging role of droxidopa. Vasc Health Risk Manag. 2014 Apr 3;10:169-76. doi: 10.2147/VHRM.S53983. eCollection 2014. PMID 24729712
- [Background] Hauser RA, Isaacson S, Lisk JP, Hewitt LA, Rowse G. Droxidopa for the short-term treatment of symptomatic neurogenic orthostatic hypotension in Parkinson's disease (nOH306B). Mov Disord. 2015 Apr 15;30(5):646-54. doi: 10.1002/mds.26086. Epub 2014 Dec 9. PMID 25487613
- [Background] Keating GM. Droxidopa: a review of its use in symptomatic neurogenic orthostatic hypotension. Drugs. 2015 Feb;75(2):197-206. doi: 10.1007/s40265-014-0342-1. PMID 25559422
- [Background] Ross AJ, Stewart JM. Prospects for droxidopa in neurogenic orthostatic hypotension. Hypertension. 2015 Jan;65(1):34-5. doi: 10.1161/HYPERTENSIONAHA.114.04204. Epub 2014 Oct 27. No abstract available. PMID 25350983
- [Background] Vijayan J, Sharma VK. Neurogenic orthostatic hypotension - management update and role of droxidopa. Ther Clin Risk Manag. 2015 Jun 8;11:915-23. doi: 10.2147/TCRM.S68439. eCollection 2015. PMID 26089676
- [Background] Isaacson S, Vernino S, Ziemann A, Rowse GJ, Kalu U, White WB. Long-term safety of droxidopa in patients with symptomatic neurogenic orthostatic hypotension. J Am Soc Hypertens. 2016 Oct;10(10):755-762. doi: 10.1016/j.jash.2016.07.010. Epub 2016 Aug 4. PMID 27614923
- [Background] Strassheim V, Newton JL, Tan MP, Frith J. Droxidopa for orthostatic hypotension: a systematic review and meta-analysis. J Hypertens. 2016 Oct;34(10):1933-41. doi: 10.1097/HJH.0000000000001043. PMID 27442791
- [Background] Freeman R, Landsberg L, Young J. The treatment of neurogenic orthostatic hypotension with 3,4-DL-threo-dihydroxyphenylserine: a randomized, placebo-controlled, crossover trial. Neurology. 1999 Dec 10;53(9):2151-7. doi: 10.1212/wnl.53.9.2151. PMID 10599797
- [Background] Zhao J, Wecht JM, Zhang Y, Wen X, Zeman R, Bauman WA, Cardozo C. iNOS expression in rat aorta is increased after spinal cord transection: a possible cause of orthostatic hypotension in man. Neurosci Lett. 2007 Mar 30;415(3):210-4. doi: 10.1016/j.neulet.2007.01.025. Epub 2007 Jan 14. PMID 17287083
- [Background] Spinal Cord Injury (SCI) 2016 Facts and Figures at a Glance. J Spinal Cord Med. 2016 Jul;39(4):493-4. doi: 10.1080/10790268.2016.1210925. No abstract available. PMID 27471859

RESULTS

PARTICIPANT FLOW:
Groups:
- Study 2: Blinded Placebo/Northera: Participants will then be administered either oral optimal dose of Northera (Droxidopa) or matching placebo in a double-blinded manner and will remain in the supine position for 60 minutes. Subjects will remain in their wheelchair for instrumentation, which will include: 1) ECG, 2) brachial BP, 3) finger arteriolar BP and 4) Cerebral Blood Flow velocity (CBFv).
  Northera: Study 1 is a dose optimization, open-label trial of Northera from a dose range of 200mg up to 800mg.
  Placebo: Study 2 is blinded placebo controlled trial using the individualized optimal dose of droxidopa determined by study 1.
- Study 2: Blinded Northera/Placebo: Participants will then be administered either oral optimal dose of Northera (Droxidopa) or matching placebo in a double-blinded manner and will remain in the supine position for 60 minutes. Subjects will remain in their wheelchair for instrumentation, which will include: 1) ECG, 2) brachial BP, 3) finger arteriolar BP and 4) Cerebral Blood Flow velocity (CBFv).
Period: Overall Study
Arm/Group | Study 1: Dose Optimization of Northera | Study 2: Blinded Placebo/Northera | Study 2: Blinded Northera/Placebo
Started | 15 | 4 | 2
Completed | 13 | 4 | 2
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study 1: Dose Optimization of Northera | Study 2: Blinded Placebo/Northera | Study 2: Blinded Northera/Placebo | Total
Number analyzed (Participants) | 13 | 4 | 2 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 2 | 19
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.54 (9.9) | 41 (13) | 37 (2) | 40.65 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 0 | 4
  Male | 9 | 4 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 11 | 1 | 1 | 13
  More than one race | 0 | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 4 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Systolic BP Within a Normotensive Range
Description: To determine the proportion (%) of normotensive systolic blood pressure for males=(110-120 mmHg); and females=(101-120 mmHg) following administration of droxidopa.
Time Frame: up to 240 minutes following administration of droxidopa
Measure: Number; unit: Systolic Blood Pressure Recordings
Units Other Than Participants: Systolic Blood Pressure Recordings
Groups:
- Study 2: Placebo; Study 2: Northera: Participants will then be administered either oral optimal dose of Northera (Droxidopa) or matching placebo in a double-blinded manner and will remain in the supine position for 60 minutes. Subjects will remain in their wheelchair for instrumentation, which will include: 1) ECG, 2) brachial BP, 3) finger arteriolar BP and 4) Cerebral Blood Flow velocity (CBFv).
Arm/Group | Study 1: Dose Optimization of Northera | Study 2: Placebo | Study 2: Northera
Number analyzed (Participants) | 15 | 6 | 6
Number analyzed (Systolic Blood Pressure Recordings) | 1282 | 412 | 402
Systolic Blood Pressure Recordings | 167 | 117 | 89

2. Secondary Outcome: Supine Systolic Blood Pressure
Description: To measure supine systolic blood pressure following administration of droxidopa compared to placebo in hypotensive participants with SCI
Time Frame: within 60 minutes of administration of droxidopa or placebo
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Study 1: Dose Optimization Northera; Study 2: Placebo: Subjects will be administered oral droxidopa in a dose escalation, open-label manner beginning with 200 mg. The dose will be adjusted upwards by 100 mg on subsequent visits until average Systolic Blood Pressure (SBP) recorded 60-120 minutes after dose administration is 111-139 mmHg in males and 101-139 mmHg in females, sustained elevation (≥ 30 consecutive minutes) in seated SBP ≥ 140/100 mmHg, maximum dose of 800 mg is reached without adequate SBP response. Subjects will visit the testing laboratory on as few as 1 (200 mg) and as many as 7 (800 mg) days. Seated cardiovascular assessments will be monitored and recorded at 15-minute intervals for 4-hours, and the side effects questionnaire will be administered hourly during the 4-hour study. Each study visit will take about 5 hours.
  Northera: Study 1 is a dose optimization, open-label trial of Northera from a dose range of 200mg up to 800mg.
- Study 2: Northera: Participants will then be administered either oral optimal dose of Northera (Droxidopa) or matching placebo in a double-blinded manner and will remain in the supine position for 60 minutes. Subjects will remain in their wheelchair for instrumentation, which will include: 1) ECG, 2) brachial BP, 3) finger arteriolar BP and 4) Cerebral Blood Flow velocity (CBFv).
  Northera: Study 1 is a dose optimization, open-label trial of Northera from a dose range of 200mg up to 800mg.
  Placebo: Study 2 is blinded placebo controlled trial using the individualized optimal dose of droxidopa determined by study 1.
Arm/Group | Study 1: Dose Optimization Northera | Study 2: Placebo | Study 2: Northera
Number analyzed (Participants) | 15 | 6 | 6
mmHg | 99.9 (12.3) | 110.9 (10.8) | 107.9 (8.7)

3. Secondary Outcome: Orthostatic Systolic Blood Pressure
Description: To document systolic blood pressure responses to head-up tilt to 70 degrees following administration of droxidopa compared to placebo in hypotensive participants with SCI.
Time Frame: 60-90 minutes following administration of droxidopa or placebo
Population: Participants did not undergo a 70 degree head-up tilt in Study 1 the dose optimization trial.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study 1: Dose Optimization Northera | Study 2: Placebo | Study 2: Northera
Number analyzed (Participants) | 0 | 6 | 6
mmHg |  | 99.92 (11.03) | 91.99 (9.85)

4. Secondary Outcome: Orthostatic Cerebral Blood Flow
Description: To compare cerebral blood flow velocity in the middle cerebral artery following administration of placebo compared to administration of Northera (Droxidopa)
Time Frame: 60-90 minutes following administration of droxidopa or placebo
Population: We did not assess middle cerebral artery cerebral blood flow velocity in Study 1 following administration of Northera
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Study 1: Dose Optimization of Northera | Study 2: Placebo | Study 2: Northera
Number analyzed (Participants) | 0 | 6 | 6
cm/sec |  | 36.4 (7.23) | 36.8 (5.26)

ADVERSE EVENTS:
Time Frame: 2 months
Description: No greater risk in SAE or mortality than typical for the study population.
Arm/Group | Study 1: Dose Optimization of Northera | Study 2: Northera | Study 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03602014/Prot_SAP_ICF_002.pdf